CLINICAL TRIAL: NCT02280512
Title: Intraoperative Monitoring With Noninvasive Near-infrared Spectroscopy and Noninvasive Cardiac Output Measurement, and Postoperative Outcome in Elderly Patients With Fractures of Lower Extremities
Brief Title: Intra-op Monitoring With NIRS and NICOM, and Surgical Outcome in Elderly Patients With Fractures of Lower Limbs
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201407114RIND
Record Dates: First submitted 2014-10-27; First posted 2014-10-31 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Femoral Fractures; Tibial Fractures
Keywords: noninvasive cardiac output measurement(NICOM); Leg fractures; Near-Infrared Spectroscopy (NIRS); Intensive care unit(ICU)
MeSH Terms: conditions — Femoral Fractures; Tibial Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- elderly with fractures: patients more than 65 years old accepting surgeries for lower extremities fracture
  Interventions: Device: elderly with fractures

INTERVENTIONS:
Device: elderly with fractures — hemodynamic monitoring with NICOM and tissue perfusion monitoring with NIRS

SUMMARY:
In Taiwan, about 75.92% of the elderlies above 65 years old suffered from chronic diseases or major diseases, especially in circulatory system. Thus, dramatic hemodynamic change is often observed in surgeries in this population. Due to osteoporosis and high-prevalence morbidities, trauma with fracture is quite common. These elderlies are more vulnerable to have complications, poor prognosis and decompensated organ functions.

The investigators would like to observe the perfusion of different tissue intra-operatively, and to find the correlation with surgical outcome. There are many non-invasive hemodynamic monitors nowadays. In our study, the investigators will use noninvasive cardiac output measurement(NICOM), and non-invasive transcutaneous near infrared spectroscopy(NIRS) to observe hemodynamic change and tissue perfusion. After the surgery, the duration in ICU will be recorded. A questionnaire, SF-36, will be mailed to the patients 2 months after the surgery to measure the psychometric status.

DETAILED DESCRIPTION:
Aging is associated with progressive loss of functional reserve in all organ systems. For most people, physiologic compensation for age-related changes is adequate. However, it is easy to decompensate under stressful circumstances, such as surgery and illness. Under the specific physiologic phenomenon, geriatric anesthesia is acquired for more intensive monitoring. In Taiwan, about 75.92% of the elderlies above 65 years old suffered from chronic diseases or major diseases, especially in circulatory system. Thus, dramatic hemodynamic change is often observed in surgeries in this population. For the elderlies with fracture are more vulnerable to have complications, poor prognosis and decompensated organ functions.

In our daily practice, the surgeries for fracture in lower extremities can performed under either general anesthesia or regional anesthesia, such as spinal anesthesia epidural anesthesia, and nerve block. The anesthetic method is determined under each patient's condition. EKG, arterial catheter, pulse oximeter are usually basic for intra-operative monitoring. However, these tools are unable to inform us the real-time cardiac output and the exact status of tissue perfusion. Nowadays, there are many non-invasive instruments able to estimate more detailed hemodynamic parameters, which are very crucial during anesthesia.1 But these instruments are not widely used in our daily practices. We need more researches to support the beneficial roles of these non-invasive monitors to high-risk patients during surgery.

Due to the hemodynamic feature in elderlies, we will use conventional measurements as EKG, arterial blood pressure and pulse oximeter. To measure the perfusion of the lower extremities, we use a relative new tool, the non-invasive transcutaneous near infrared spectroscopy (NIRS).2,3 NIRS was used as the cerebral oximetry to measure the tissue perfusion of the cerebral cortex. It uses reflectance oximetry to measure the oxygen saturation of the tissue underneath the sensor.1 Recently, NIRS has been proved not only to continuously monitor tissue oxygenation saturation (StO2) continuously, but also to predict the patient's poor prognosis.3,4 To measure the cardiac output intra-operatively, we will use the non-invasive cardiac output monitor (NICOM®, Cheetah). Bioreactance technique allows the measurement of hemodynamic changes via four electrodes placed on the thorax. The electrical current crossing the thorax makes "signal phase shift", which is related to changes in the volume of the thoracic aorta. Thus, the volume change in the thoracic aorta is able to estimate stroke volume.1,5 Postoperative prognosis is adjusted with the recovery of ambulation, the duration of ICU stay, the morbidity and mortality, and the questionnaire (SF-36) about quality of life.

ELIGIBILITY:
Inclusion criteria:

* Patients more than 65 years old accepting surgeries for lower extremities fracture

Exclusion criteria:

* Skin lesions over the sites where NIRS patches and NICOM electrodes are about to be attached.
* Patients with history of being allergic to NIRS patches or NICOM electrodes.
* Patients with pleural effusion or pericardial effusion.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patient older than 65 years old with fractures of lower limbs
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Psychometric status in 3 months after the surgery | 3 months
  Evaluation via questionnaire, SF-36

SECONDARY OUTCOMES:
ICU stay | 2 Days
  If the patient was admitted to intensive care units(ICU) after the operation, the duration of staying in ICU is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Po-Yuan Shih, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan